CLINICAL TRIAL: NCT07212270
Title: Effectiveness of Intraseptal Anesthesia for Periodontal Surgical Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Natasa Nikolic Jakoba, professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBelgrade 36/8 (2)
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Periodontitis; Gingivitis and Periodontal Diseases
MeSH Terms: conditions — Periodontitis; Gingivitis; Periodontal Diseases | interventions — Gingivectomy; Gingivoplasty

STUDY DESIGN:
Intervention Model Description: 2 parallel groups, each with the experimental and the control group
Who Masked: Care Provider
Masking Description: Periodontist do not know the type of anesthesia given by the investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GG test (Experimental): Patient subjected to gingivectomy and gingivoplasty interventions and anesthesia of choice is intraseptal anesthesia.
  Interventions: Procedure: gingivectomy and gingivoplasty
- GG control (Active Comparator): Patient subjected to gingivectomy and gingivoplasty interventions under the local infiltration anesthesia.
  Interventions: Procedure: gingivectomy and gingivoplasty
- PF test (Experimental): Patients undergoing periodontal flap surgery under the intraseptal anesthesia.
  Interventions: Procedure: periodontal flap surgery
- PF control (Active Comparator): Patients undergoing periodontal flap surgery under the local infiltration anesthesia.
  Interventions: Procedure: periodontal flap surgery

INTERVENTIONS:
Procedure: periodontal flap surgery — Open flap debridement with intra-sulcular incisions or flaps with para-marginal incisions were performed by lifting the mucoperiosteal flap and debriding the periodontal defect under visual control.
  Arms: PF control; PF test
Procedure: gingivectomy and gingivoplasty — surgical methods for the excision of hyperplastically enlarged gingiva.
  Arms: GG control; GG test

SUMMARY:
The primary aim of this study is to evaluate the efficacy of intraseptal anesthesia using 0.3 mL of 4% articaine with 1:100,000 epinephrine (4% Ar+Ep) for periodontal flap surgery in patients with periodontitis and for gingivectomy/ gingivoplasty for the excision of hyperplastic gingival enlargements. The secondary aim is to compare clinical anesthetic parameters between the ISA and conventional anesthesia techniques.

DETAILED DESCRIPTION:
In the test groups every patient is going to receive injections of 0.3 mL of 4% articaine with 1: 100,000 epinephrine (ORABLOC ® , 40 mg/ml Articaine + 0.01 mg/ml Epinephrine, PIERREL S.P.A, Capua, Italy), with a computer controlled anesthesia delivery system (Anaeject®, Septodont, Sallanches, France). In the control groups all surgical procedures is going to be performed under infiltration anesthesia, as commonly used in periodontal surgery. The success rate and the anesthetic field widths is going to be recorded by pinprick testing. The pain levels will be recorded using the Visual Analogue Scale (VAS) for the administration of anesthesia, during the surgical procedure and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years good systemic health
* gingivitis or periodontitis stage II and III
* at least 20 teeth present.

Exclusion Criteria:

* allergy to 4%Ar+Ep
* pregnant or lactating females
* medication uptake and diseases affecting the periodontal tissues
* acute pain, swelling, and presence of gingival lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The anesthetic efficacy | 5 min after injection
  The absence of pain for two pinprick tests in a row.
The width of the anesthetic field on the buccal side | 5 min after injection
  maximal distance between the two painless needle's pricks on the buccal aspect of attached gingiva
The width of the anesthetic field on oral side | 5 min after injection
  The maximal distance between the two painless needle's pricks on the oral aspect of the attached gingiva.
VASa | immediately after anesthetic administration
  The intensity of pain measured on 100mm Visual Analogue Scale, where 0 represented no pain and 100 the worst pain imaginable.
VASi | at the end of the treatment
  The intensity of pain measured on 100mm Visual Analogue Scale, where 0 represented no pain and 100 the worst pain imaginable.
VASp | one day follow-up
  The intensity of pain measured on 100mm Visual Analogue Scale, where 0 represented no pain and 100 the worst pain imaginable.
The duration | form start to finish od intervention
  The duration of intervention, measured in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology and Oral medicine, School of Dental Medicine, University of Belgrade, Belgrade, Serbia